CLINICAL TRIAL: NCT00804999
Title: Two Phase Clinical Study of the Impact of Contact Lenses and Solutions on Corneal Structure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Christine Sindt (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Sponsor-Investigator, Christine Sindt, Principal Investigator, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 200806729
Record Dates: First submitted 2008-12-05; First posted 2008-12-09 (Estimated); Results first posted 2018-01-23 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2017-12

CONDITIONS: Normal Contact Lens Wear
Keywords: confocal microscopy; contact lens wear; contact lens solutions; sodium fluorescein

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo 1 (Placebo Comparator): Subjects that have never worn contacts with no ocular problems were selected. A baseline HRT was performed. Trial contact lenses were soaked in clear care solution for 10 hours. After 10 hours of the lenses soaking in clear care the subject returned. The contacts lenses that were soaked in clear care were inserted onto the patients eyes. The patient then wore the contacts for two hours. After two hours the contact lenses were removed. An HRT was performed immediately after removing the contact lenses. The HRT scans were analyzed for dendritic cell migration, basal cell epithelial density and nerve density and tortuosity.
  Interventions: Drug: Clear Care
- Renu (Active Comparator): Subjects that had worn contacts for at least two weeks without incident were selected. A baseline HRT was performed.Trial contacts lenses were soaked in ReNu contact solution for 10 hours. After 10 hours of the lenses soaking in ReNu the subject returned. The contacts were inserted onto the patients eyes. The patient then wore the contacts for two hours. After two hours the contacts lenses were removed. An HRT both with and without sodium fluorescein was performed immediately after removing the contact lenses.The HRT scans were analyzed for dendritic cell migration, basal cell epithelial density and nerve density and tortuosity.
  Interventions: Drug: ReNu
- Optifree (Active Comparator): Subjects that had worn contacts for at least two weeks without incident were selected. A baseline HRT was performed.Trial contacts lenses were soaked in Optifree Replenish contact solution for 10 hours. After 10 hours of the lenses soaking in Optifree Replenish the subject returned. The contacts were inserted onto the patients eyes. The patient wore contacts the for two hours. After two hours the contacts were removed. An HRT both with and without sodium fluorescein was performed immediately after removing the contact lenses.The HRT scans were analyzed for dendritic cell migration, basal cell epithelial density and nerve density and tortuosity.
  Interventions: Drug: OPTI-FREE

INTERVENTIONS:
Drug: Clear Care — neutralized Clear Care
  Other Names: hydrogen peroxide disinfecting solution
  Arms: Placebo 1
Drug: ReNu — overnight soak in solution
  Arms: Renu
Drug: OPTI-FREE — overnight soak in solution
  Other Names: Replenish
  Arms: Optifree

SUMMARY:
Assess the usefulness of using confocal microscopy to examine changes to the structure of the cornea and to identify any potential consequences of contact lens wear and/or solution use.

DETAILED DESCRIPTION:
Several types of solutions are used in contact lens wear.

Each contact lens solution used to disinfect contacts have different ingredients even though they all disinfect the contacts.

The objective of this study is to examine the layers of the cornea via HRT in order to assess the usefulness of this technology and to identify any potential consequences of contact lens wear and/or care solution used.

ELIGIBILITY:
Inclusion Criteria:

* Vision correctable to 20/30 or better in both eyes
* Successful soft contact lens wear for at least 2 weeks prior to enrollment

Exclusion Criteria:

* History of hypersensitivity to any of the components in any of the lens solutions
* One functional eye or a monofit lens
* Any abnormal slit-lamp finding at baseline
* Use of topical ocular meds
* Any systemic condition with significant ocular side effects or that interfere with contact lens wear
* Enrollment of the investigator's office staff, relatives or members of their respective households
* Enrollment of more than one member of the same household

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2008-11-01 (Actual); Primary Completion 2009-03-01 (Actual); Study Completion 2009-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine W Sindt, O.D., Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Contact Lens Clinic, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD.

REFERENCES:
- [Background] Patel DV, McGhee CN. In vivo laser scanning confocal microscopy confirms that the human corneal sub-basal nerve plexus is a highly dynamic structure. Invest Ophthalmol Vis Sci. 2008 Aug;49(8):3409-12. doi: 10.1167/iovs.08-1951. Epub 2008 Apr 25. PMID 18441297
- [Background] Dosso AA, Rungger-Brandle E. Clinical course of epidemic keratoconjunctivitis: evaluation by in vivo confocal microscopy. Cornea. 2008 Apr;27(3):263-8. doi: 10.1097/ICO.0b013e31815b7d7d. PMID 18362649
- [Background] Fonn D, Simpson T, Woods J, Woods C. New technologies to assess lens-mediated effects of the cornea. Eye Contact Lens. 2007 Nov;33(6 Pt 2):364-70; discussion 382. doi: 10.1097/ICL.0b013e318157c98f. PMID 17975422
- [Background] Bantseev V, McCanna DJ, Driot JY, Ward KW, Sivak JG. Biocompatibility of contact lens solutions using confocal laser scanning microscopy and the in vitro bovine cornea. Eye Contact Lens. 2007 Nov;33(6 Pt 1):308-16. doi: 10.1097/ICL.0b013e31803c55ad. PMID 17993827
- [Background] Kanavi MR, Javadi M, Yazdani S, Mirdehghanm S. Sensitivity and specificity of confocal scan in the diagnosis of infectious keratitis. Cornea. 2007 Aug;26(7):782-6. doi: 10.1097/ICO.0b013e318064582d. PMID 17667609
- [Background] Efron N. Contact lens-induced changes in the anterior eye as observed in vivo with the confocal microscope. Prog Retin Eye Res. 2007 Jul;26(4):398-436. doi: 10.1016/j.preteyeres.2007.03.003. Epub 2007 Apr 1. PMID 17498998
- [Background] Zhivov A, Stave J, Vollmar B, Guthoff R. In vivo confocal microscopic evaluation of langerhans cell density and distribution in the corneal epithelium of healthy volunteers and contact lens wearers. Cornea. 2007 Jan;26(1):47-54. doi: 10.1097/ICO.0b013e31802e3b55. PMID 17198013
- [Background] Bastion ML, Mohamad MH. Study of the factors associated with the presence of white dots in the corneas of regular soft contact lens users from an Asian country. Eye Contact Lens. 2006 Sep;32(5):223-7. doi: 10.1097/01.icl.0000199891.35160.68. PMID 16974154
- [Background] Su PY, Hu FR, Chen YM, Han JH, Chen WL. Dendritiform cells found in central cornea by in-vivo confocal microscopy in a patient with mixed bacterial keratitis. Ocul Immunol Inflamm. 2006 Aug;14(4):241-4. doi: 10.1080/09273940600732398. PMID 16911987
- [Background] Nguyen TH, Dudek LT, Krisciunas TC, Matiaco P, Planck SR, Mathers WD, Rosenbaum JT. In vivo confocal microscopy: increased conjunctival or episcleral leukocyte adhesion in patients who wear contact lenses with lower oxygen permeability (Dk) values. Cornea. 2004 Oct;23(7):695-700. doi: 10.1097/01.ico.0000127482.00843.c8. PMID 15448495
- [Background] Patel SV, McLaren JW, Hodge DO, Bourne WM. Confocal microscopy in vivo in corneas of long-term contact lens wearers. Invest Ophthalmol Vis Sci. 2002 Apr;43(4):995-1003. PMID 11923239

RESULTS

PARTICIPANT FLOW:
Groups:
- Non Contact Wearer Using Clear Care: neutralized Clear Care and no contact lens wear
  Clear Care: neutralized Clear Care
- Overnight Soaking With Renu: ReNu with and without sodium fluorescein
  ReNu MultiPlus MPS: overnight soak in solution
- Overnight Soak in Optifree: RepleniSH with and without sodium fluorescein
  ReNu MultiPlus MPS: overnight soak in solution
  OPTI-FREE RepleniSH MPDS: overnight soak in solution
- Overnight Soak in Optifree Replnish: ReNu and RepleniSH
  OPTI-FREE RepleniSH MPDS: overnight soak in solution
Period: Overall Study
Arm/Group | Non Contact Wearer Using Clear Care | Overnight Soaking With Renu | Overnight Soak in Optifree | Overnight Soak in Optifree Replnish
Started | 15 | 12 | 14 | 10
Completed | 15 | 12 | 14 | 10
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Non Contact Lens Wearers Using Clear Care: neutralized Clear Care and no contact lens wear
  Clear Care: neutralized Clear Care
- Overnight Soaking in Optifree: RepleniSH with and without sodium fluorescein
  ReNu MultiPlus MPS: overnight soak in solution
  OPTI-FREE RepleniSH MPDS: overnight soak in solution
- Overnight Soaking in Optifree Replinish: ReNu and RepleniSH
  OPTI-FREE RepleniSH MPDS: overnight soak in solution
- Total: Total of all reporting groups
Arm/Group | Non Contact Lens Wearers Using Clear Care | Overnight Soaking With Renu | Overnight Soaking in Optifree | Overnight Soaking in Optifree Replinish | Total
Number analyzed (Participants) | 15 | 12 | 14 | 10 | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 15 | 12 | 14 | 10 | 51
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 11 | 13 | 9 | 46
  Male | 2 | 1 | 1 | 1 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 12 | 14 | 10 | 51

OUTCOME MEASURES:

1. Primary Outcome: HRT Corneal Scan
Description: Looking for cell density
Time Frame: baseline and 2 hours
Measure: Mean (Standard Deviation); unit: cells/mm^3
Groups:
- Non Contact Wearing Using Clear Care: neutralized Clear Care and no contact lens wear
  Clear Care: neutralized Clear Care
Arm/Group | Non Contact Wearing Using Clear Care | Overnight Soaking With Renu | Overnight Soaking in Optifree | Overnight Soaking in Optifree Replinish
Number analyzed (Participants) | 15 | 12 | 14 | 10
cells/mm^3
  Baseline | 85 (112) | 66 (44) | 49 (28) | 63 (081)
  Two hours | 87 (110) | 65 (48) | 51 (32) | 61 (77)

ADVERSE EVENTS:
Time Frame: 3 weeks
Arm/Group | Non Contact Wearing Using Clear Care | Overnight Soaking With Renu | Overnight Soaking in Optifree | Overnight Soaking in Optifree Replinish
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/12 | 0/14 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/12 | 0/14 | 0/10
Other Adverse Events (participants affected / at risk) | 0/15 | 0/12 | 0/14 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No